CLINICAL TRIAL: NCT03973138
Title: Visual Outcomes and the Predictive Factors in Chinese Patients With Diabetic Macular Edema Treated With Ranibizumab
Acronym: IVRDME
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZOC-IVRDME02
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Diabetic Macular Edema
Keywords: Macular edema; ranibizumab; Mpredictive factor
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): DME patients who were diagnosed through fundus manifestations and FFA examination were treated by intravitreal injections of ranibizumab under the pro re nata (PRN) treatment regimen.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — DME patients who were diagnosed through fundus manifestations and FFA examination were treated by intravitreal injections of ranibizumab (0.5mg Lucentis®; Genentech, South San Francisco, CA) under the pro re nata (PRN) treatment regimen. The retreatment were conducted if BCVA was reduced by 0.1 logarithm of the minimal angle of resolution (logMAR) value or more from maximum acuity or if OCT central subfield thickness was more than 300μm.

SUMMARY:
The aim of this study is to evaluate the one-year visual outcome and prognostic factors after intraocular injections of ranibizumab under pro re nata treatment regimen for the patients with diabetic macular edema (DME).

DETAILED DESCRIPTION:
The aim of this study is to evaluate the one-year visual outcome and prognostic factors after intraocular injections of ranibizumab under pro re nata treatment regimen for the patients with diabetic macular edema (DME). Mean change of logarithm of the minimal angle of resolution (logMAR) visual acuity (VA), central foveal thickness (CFT), as well as predictive factors including best-corrected visual acuity (BCVA) were assessed.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients (aged>18 years) with DME who had a best-corrected visual acuity (BCVA) between 20/32 and 20/200, and CRT≥300μm; 2) clinically significant DME confirmed by both fundus fluorescein angiography (FFA) and optical coherence tomography (OCT) (Spectralis HRA+OCT; Heidelberg Engineering, Germany); 3) decreased vision caused by foveal thickening from DME, which could not be explained by any other cause.

Exclusion Criteria:

* 1) previous anti-VEGF or laser treatment; 2) proliferative diabetic retinopathy who required immediate panretinal photocoagulation; 3) active proliferative diabetic retinopathy; 4) other causes for macular edema, for example, branch retinal vein occlusion; 5) other causes of visual loss in the study; 6) unstable systemic conditions, for example, uncontrolled blood pressure, stroke, renal or kidney failure.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity | one year
  changes of best-corrected visual acuity

SECONDARY OUTCOMES:
Central foveal thickness | one year
  changes of central foveal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Kunbei Lai, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lai K, Huang C, Li L, Gong Y, Xu F, Zhong X, Lu L, Jin C. Anatomical and functional responses in eyes with diabetic macular edema treated with "1 + PRN" ranibizumab: one-year outcomes in population of mainland China. BMC Ophthalmol. 2020 Jun 15;20(1):229. doi: 10.1186/s12886-020-01510-0. PMID 32539744